# Study Protocol: Mindfulness-Based Childbirth and Parenting Education

#### 1. Introduction

Date of Last Revision: July 30, 2025

## 2. Objectives

Primary Objective:

• To examine the effect of the mindfulness-based education program on prenatal distress levels, measured using the Tilburg Pregnancy Distress Scale (TPDS).

#### Secondary Objectives:

 To assess the impact on mindful awareness (MAAS), fear of childbirth (W-DEQ), and maternal attachment.

## 3. Methodology

This randomized controlled trial included 31 pregnant women aged 18 to 35. Participants were randomly assigned to the intervention group (n=16) or the control group (n=15). The intervention group received an 8-week online MBCP-based training. The control group received standard prenatal care.

#### 4. Intervention

The intervention included weekly 120-minute online sessions comprising formal mindfulness practices (e.g., body scan, mindful breathing), informal mindfulness practices (e.g., mindful eating), psychoeducation, and group reflection. Participants also completed daily home practice with guided audio recordings.

#### **5. Outcome Measures**

**Primary Outcome:** 

• - Change in prenatal distress scores (TPDS) from baseline to post-intervention.

### **Secondary Outcomes:**

• - Changes in mindful awareness (MAAS), fear of childbirth (W-DEQ), and maternal attachment measured postpartum.

#### 6. Eligibility Criteria

Inclusion Criteria:

- - Pregnant women aged 18–35
- - TPDS score ≥ 28
- - Gestational age between 24–32 weeks

- - First-time pregnancy
- - Able to attend online sessions

#### Exclusion Criteria:

- - High-risk pregnancies or multiple gestation
- - Prior mindfulness training
- - Major psychiatric or medical conditions

### 7. Ethics and Consent

The study was approved by the Institutional Review Board. Written informed consent was obtained from all participants.

Date: August 7, 2025

Principal Investigator: Merve Gül Tiren

Mindfulness-Based Childbirth and Parenting Education Study Protocol